CLINICAL TRIAL: NCT00466102
Title: RADAR: A Randomized Discontinuation Phase II Study to Determine the Efficacy of RAD001 in Breast Cancer Patients With Bone Metastases
Brief Title: Efficacy of RAD001 in Breast Cancer Patients With Bone Metastases
Acronym: RADAR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GBG 41
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Bone metastases as only metastatic site; Breast cancer, HER2 negative; Bone metastasis as only metastatic site; Pretreated with endocrine therapy; Up to one previous chemotherapy; Previous treatment with bisphosphonates allowed
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Patients with stable disease after 8 week run in randomized to RAD001 (blinded)
  Interventions: Drug: RAD001
- 2 (Placebo Comparator): Patients with stable disease after 8 week run in receive placebo (blinded)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RAD001 — Tablet of 5 mg, 2 tablets (10 mg) are taken once daily during study therapy
  Arms: 1
Drug: Placebo — 2 tablets are taken once daily during study therapy
  Arms: 2

SUMMARY:
The purpose of this study is to determine wether RAD001 can inhibit growth of tumour cells and/or stop the formation and activity of bone degrading osteoclasts.

DETAILED DESCRIPTION:
RAD001 is an orally bioavailable and well tolerated rapamycin ester analogue, which acts by selectively inhibiting mTOR (mammalian target of rapamycin). mTor is an intracellular protein kinase implicated in the control of cellular proliferation in neoplastic cells. Treatment with RAD001 has been shown to inhibit these signalling events and leads to growth retardation of tumour cells. In addition RAD001 in vitro stops the formation and activity of osteoclasts. Therefore a therapy of advanced breast cancer with progressive bone metastases seems to be reasonable with RAD001.

Comparison:

All patients receive RAD001 in an 8 week run in phase. Patients who show a response after 8 weeks will continue receiving RAD001. All patients with stable disease after the run in phase will be randomised to receive either RAD001 or placebo and will be followed up until progression of disease. Patients with progressive disease after the 8 week run in phase will be withdrawn from the trial.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirements.
* Histologically confirmed invasive adenocarcinoma of the breast.
* Primary tumour or metastasis negative or positive (≥ 10% positive stained cells) for oestrogen and/or progesterone receptor detected by immunohistochemistry.
* Single or multiple bone metastasis (x-ray, CT or MRI) as only metastatic site.
* Postmenopausal hormone receptor positive patients should have received an aromatase inhibitor in any given previous breast cancer therapy. Concurrent endocrine treatment for metastatic bone disease is obligatory. Previous treatment with bisphosphonates is allowed.
* Up to one previous chemotherapy for metastatic disease is allowed.
* Patients must have either measurable or non-measurable target lesions according to the WHO criteria.
* At least 1 target lesion must be completely outside the radiation portal or there must be pathologic proof of progressive disease.
* At least 2 weeks since major surgery with full recovery.
* Complete staging within 4 weeks prior to registration.
* Karnofsky performance status evaluation > 60%.
* Age >18 years.
* Absolute neutrophil count >1,500 cells/µl, platelet count >100,000 cells/µl.
* Bilirubin >1.5x the upper normal limit for the institution (UNL); elevation of transaminases, alkaline phosphatase < 2.5x UNL and serum albumin < 30g/l. Normal renal function (creatinine >1.5x upper normal limit)
* If of childbearing potential, negative pregnancy test. In addition the patient has to agree to use an effective method to avoid pregnancy for the duration of the study.

Exclusion Criteria:

* Known hypersensitivity reaction to the compounds or incorporated substances (e.g. everolimus or sirolimus [rapamycin] or lactose).
* Concurrent immunotherapy or hormone replacement therapy and use of hormonal contraceptives.
* Need for chemotherapy or irradiation of bone metastasis during study treatment
* HER2 positive primary tumour and/or lesion
* Evidence of metastasis in other organs
* Uncompensated diabetes mellitus; fasting value of blood sugar of >120 (mg/dl)
* Corrected (adjusted for serum albumin) serum calcium concentration < 8.0 mg/dl (2.00 mmol/l) or > 12.0 mg/dl (3.00 mmol/l)
* Abnormal renal function as evidenced by a calculated creatinine clearance < 30 ml/minute
* Life expectancy of less than 3 months
* Serious intercurrent medical or psychiatric illness that may interfere with the planned treatment (including AIDS and serious active infection).
* History of other malignancy within the last 5 years which could affect the diagnosis or assessment of metastatic breast cancer
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry.
* Patients being treated with drugs recognized as being strong inhibitors or inducers of the isoenzyme CYP3A (e.g. rifabutin, rifampicin, clarithromycin, ketoconazole, itraconazole, ritonavir, telithromycin, erythromycin, verapamil, dilitazem) within the last 5 days or the expected need for these treatments during study participation.
* Pregnant or nursing women.
* The patient is not accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre which could be the Principal or Co-Investigator's site.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2006-12; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To determine the time to progression (TTP) in patients with no change in bone metastases after an 8 week run in treatment with RAD001 compared to placebo | 40 weeks

SECONDARY OUTCOMES:
To determine the objective response rate after 8 weeks of RAD001 | 8 weeks
To determine the TTP in patients with a response after 8 weeks of RAD001 | 8 weeks
To determine the overall clinical benefit defined as CR, PR or stable disease > 24 weeks for patients continuing RAD001 after the 8 week run in phase | 40 weeks
To evaluate the safety and toxicity of RAD001 | 40 weeks
To assess the frequency of bone related events | 40 weeks
To assess changes of pain intensity during treatment | 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Maass, MD, Prof., Principal Investigator — Universitätsfrauenklinik Aachen
Locations (1):
- Dr. med. Christoph Mundhenke, Kiel, Schleswig-Holstein, Germany

REFERENCES:
- See also: Related Info — http://www.germanbreastgroup.de